CLINICAL TRIAL: NCT02715895
Title: A Clinical Trial of Infant Formula-fed
Brief Title: Clinical Trial of Infant Formula-fed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maternal and Child Health Care Hospital of Hainan Province (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CJEBP-01
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-03

CONDITIONS: Body Weight Changes
Keywords: Infant; Growth; Body Weight Changes; Infant Formula; Randomized Controlled Trial
MeSH Terms: conditions — Body Weight Changes | interventions — Milk, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Friso (Experimental): Friso formula feeding
  Interventions: Dietary Supplement: Friso
- Wyeth (Experimental): Wyeth formula feeding
  Interventions: Dietary Supplement: Wyeth
- Breast milk (Active Comparator): Breast milk feeding
  Interventions: Dietary Supplement: Breast milk

INTERVENTIONS:
Dietary Supplement: Friso — Friso formula feeding on demand for 3 months
  Arms: Friso
Dietary Supplement: Wyeth — Wyeth formula feeding on demand for 3 months
  Arms: Wyeth
Dietary Supplement: Breast milk — Breast milk feeding on demand
  Arms: Breast milk

SUMMARY:
Compared with breast milk and another commercially available formula, infants' growth rate after 12 weeks' Friso formula with different ways of processing feeding will be assessed.

DETAILED DESCRIPTION:
1. Sample size：Seventy two cases will be enrolled in breast milk group, 144 cases in formula milk group, 72 cases each in commercially available formula subgroup and Friso formula subgroup with 36 cases each in every hospital (18 male infants and 18 female infants).
2. Observation period：Observational period will maintain 12 weeks. Infants of breast milk group are fed with breast milk before inclusion and during the trial process. In the formula milk groups, if subjects were fed with other formula instead of commercially available formula and Friso formula before inclusion, then a wash-out period of no more than 2 weeks is necessary.
3. Random method: In commercially available formula subgroup and Friso formula subgroup, infants will be included randomly. Random allocation sequence is generated in six trial centers by the editorial department of Chinese Journal of Evidence-Based Pediatrics, included infants are chosen and their information including name, gender, their parents' name and telephone is reported to the editorial department of Chinese Journal of Evidence-Based Pediatrics via WeChat. Then group division information is acquired, the tested commercially available formula and Friso formula are given out to infants accordingly.
4. Match of the breast milk group: Infants with purely breast milk-fed will be chosen. Infants'gender and body weight (±5%) of breast matched with milk-fed group commercially available formula subgroup and Friso formula subgroup.
5. Blinding method: Subjects, doctors and nurses know which formula is given. Personals in charge of assessing stool character and ery secretion, and data analysis, are blind to the information of group division.
6. Data records, monitoring and management 6.1 Data records 6.1.1 Original records: Subjects' follow-up care cards are original files in this clinical trial which is in duplicate copies. One copy should be saved in hospital. Original records shall be traceable. Each researcher must strictly follow the principle of GCP and ensure that he will record any observation and discovery in the follow-up care card and case report form (CRF), all data are consistent, no optional changes are allowed. If any correction is needed, the original record must not be changed, researchers can only add extra descriptions and explain the reason, the correction needs to be signed and dated by researchers who make it.

   6.1.2 Case report form(CRF): Each in triplicate, it will be delivered to sponsors, main institutions of clinical research and participating institutions of clinical research. According to the principle of GCP, subjects' name should not appear in order to ensure their privacy. Subjects' name must be filled in the initials.

   All of the choices"□" will be marked"×". If some inspection items are not examined or missed for some reason, it should be filled in: not examined. If the specific formula dosage is unknown, it should be filled in: unknown. When filled in the numbers, it should be filled in all □. If digits are not enough, it should be filled on right side. If left side is empty, it should be filled by 0. No null terms or missing items are allowed. Researchers must ensure that all data must be consistent with the original record.

   If modifying, researchers should draw a horizontal line in the middle of the original record text, sidenote to modify, and then sign the modifier's name and the date. He must not smear or cover the original record.

   6.1.3 Data Record of subjects' guardian: It should be recorded according to the items and their definitions in the designed CRF chart.

   6.1.4 Extremum principles: The data, deviating significantly or outside the acceptable range clinically, must be verified. Clinical doctors must make the necessary instructions.

   6.1.5 Data registration and preservation: Every time after the follow-up visit, researchers should record the required information in the case report sheet timely. After the end of each subjects' observed period, researchers should accurately record relevant information from original records in the form of data in the CRF within 7 days. CRF, informed consent and other documents should be examined and signed by the project leader, then saved in the archive office of institution. If a problem is found, it should be timely dealt with and recorded.

   6.2 Data monitoring Editorial Board of Chinese Journal of Evidence-Based Pediatrics will be in charge of data monitoring of the clinical trial. CJEBP will provide data monitoring of the clinical trial to FrieslandCampina regularly in at middle experiment stage and later experiment stage. During the trial, CJEBP will investigate 6 research centers for their quality of practice at least one time, without any announcement in advance. The monitoring subjects include child care doctors, nurses and guardians of subjects enrolled in this trial.

   6.2.1 Child care doctors: monitor the quality of explaining the research to subjects' guardians and the informed consent signing; Random of distribution; The accurate measurement of body length, weight and head-circumference; judgement of gut intolerance; record of stool frequency, pictures of stools and eye secretions.

   6.2.2 Nurses: motor the accuracy of the measuring equipment; the correctness of the measuring method; the rightness of data recording (mean value of 2 measurements); the management of trial formula (reception time, check-up, distribution subjects, date and signature, recycling subjects, date, quantity of the rest formula and signature).

   6.2.3 Guardians of subjects enrolled in this trial: randomly inspect 1-2 guardians, investigate whether mixed feeding or mixed with other brand formula feeding exists; the usage of trial formula; regularity of follow-up visits; taking photos of fresh stools and eye secretions.

   6.3 Data management 6.3.1 Buildup, test and data entry of WeChat client: According to the project of the CRF，administrators will establish WeChat client, test and modify this client, and enter data after ensuring the accuracy of this client. Every researcher in each hospital uploads the measured data to administrators by WeChat client on the day he completes one case observation and measurement. In order to ensure the accuracy of the data, administrators should compare data uploaded by WeChat client with the original CRF. Subjects' guardians will upload photos of stool character and eye secretion to administrators by WeChat client at 3 points of follow-up time.

   6.3.2 Generation and correction of doubt, quality control(QC) and database shutdown: After completing data input and comparison, data administrators will verify the reliability, integrity and accuracy of data according to requirements of clinical trial scheme. If he finds loss of content or logic contradiction or filling in wrong or uncertain data, clinical monitors will send it to clinical trial centers in the form of data question table (DQF). Researchers will give answers to questions as soon as possible and reply. Data administrators will modify, confirm and correct data according to researchers' answers. After solving all of problems, quality control personnels will check the quality of database according to QC plan. Then he will close the database after check.

   6.3.3 Data check, lock and transmit blindly: Data administrators submit data management reports, and require a meeting about data-check blindly attended by principal investigator, statistical analyst, data administrators, monitors, and sponsors. Check data blindly, sign blindly data-check resolution after meeting, lock in the database; locked data will be analyzed by personnels of statistical analysis.
7. Statistic analysis 7.1 General principles: All of the statistical tests must be two-sided tests, P<0.05 is considered to be statistically significant difference for all tests. Mean, median, standard deviation, maximum, minimum, 25% and 75% quintile are used for statistical description of measurement data. Count data or level data is described by frequency ( percentage).

   SAS9.1.3 statistical software is used for statistical analysis. 7.2 Analysis of missing cases: List cases number of inclusion, completion and falling off. Loss rate and comparison between groups should be analyzed by Chi-square test and Fisher's exact probability method.

   7.3 Evaluation of effectiveness: Measurement data of indexes(Growth rate of height, weight and head circumference at 4,8,12 week, defication frequency) should be analyzed by normality test firstly. If data conforms to normal distribution, the comparation between formula milk group (commercially available formula subgroup and Friso formula subgroup) and breast milk group should be analysed by One-Way ANOVA method. LSD method is used for multiple comparisons. If data does not conform to normal distribution, then Wilcoxon Rank-Sum test is used. A level of significance is α=0.05 (two-tailed). Frequency data of indexes ( incidence of constipation at 4,8,12 week, eyes secretion) is recorded as cases or percentage. If theoretical frequency <5 or total observed frequency <30, Fisher's exact probability method is used; otherwise Chi-square test is used. A level of significance is α=0.05 (two-tailed).
8. Quality control Standardized operation procedures should be established in all of research process.

   8.1 Qualification of research institution: Research institution must be community health service centers qualified for baby healthy check-up.

   8.2 Qualification of researchers: The researchers need GCP training and work under the guidance of senior professionals.

   8.3 Trial quality control measures: ①Before the start of clinical trials, researchers (including nurses) must receive training for measurement of height, weight and head circumference; ②check measurement bed before measurement everyday. Researchers must compare scale on plastic flexible rule with that on standard steel rule and change plastic flexible if error >0.1cm. ③The pictures of the feces and eyes will be independently scored by 2 specialists under the condition of unknowing the group. ④The specialist must be responsible for experimental formula, counter locked, storage at room temperature away from light. The remaining experimental formula will be stored separately, registering number. At the end of trial, the remaining experimental formula will be sent back to sponsor.⑤Monitor: Monitor will be appointed by sponsor, ensuring subjects' interests during period of trial. Trial record and data report must be true, accurate, complete and correct, ensuring that trial must comply with both approved plan and Relevant laws.
9. Definition and management of adverse events 9.1 Definition of adverse events: adverse events are defined as those occur after a patient or a subject in a clinical study receives a tested product, the event does not necessarily have a causal relationship with the test products. Adverse events are the diseases or signs or symptoms that occur during the course of the study (including abnormal laboratory findings). Adverse events can be serious or not serious, may or may not cause the subjects to withdraw from the study. All adverse events must be recorded, and the relationship between the product and the product is evaluated.

9.2 Information collection of adverse events: researchers must know and record the following information concerning adverse events: subjects and date, description of the event, source of report, the suspected products, continuous time, frequency, extent, severity, measures taken, results and complications, the relationship with tested products.

9.3 Extent of adverse events: Mild: symptoms were not obvious, only slightly harmful to health. Middle: the symptoms are obvious, but can be tolerated, without immediate treatment. Serious: it is hard to bear.

9.4 Severity of adverse events: Serious adverse events refer to the follwing adverse events which appear at any of the dosage: leading to death, threatening life , need to be hospitalized or hospitalization has been prolonged, resulting in permanent or significant disability and loss of function, congenital anomalies or birth defects, or other significant medical events. Not serious: Those events can not be defined as serious adverse events are not serious events.

9.5 Unexpected or expected serious adverse events: Researchers must assess whether the adverse events be expected to occur or not. Expectation is evaluated by Safety Officer Medical which base on the current knowledge and existing product information. An unexpected adverse event is one that the nature, severity, frequency are inconsistent with conditions of the study and ( or) product information.

All suspected adverse events related to the tested products, as well as serious adverse events that are not expected to be serious are considered to be SUSARs (suspicious unexpected serious adverse event). SUSAR need to be reported to the management authority or independent ethics committee in a very short time.

According to the Chinese food and Drug Administration report of adverse reactions and and regulations of drug supervision, any new or serious adverse reactions of any drug must be reported within 15 days, any deaths must be reported immediately. Fax: +86-10-67184591, Email: report@adr.gov.cn.

9.6 Relationship with the tested product: Medical institutions will evaluate the relationship between adverse events and the tested product according to the following standards. ① unrelevant: there is evidence proving that adverse events are caused by other reasons. For example, adverse events are obviously caused by the disease, adverse events are consistant with effects or adverse reactions of the drugs, or adverse events had already existed before using the tested product research. ② Not likely to be relevant: it seems to have a time-relationship with the use of tested product, but the occurrence of adverse events can be explained by other reasons. ③Probably relevant: it seems to have a time-relationship with the use of tested product, and adverse events seem to have a causal relationship with the product. ④ Surely relevant: it seems to have a time-relationship with the use of tested product, and no other reasons can explain the occurrence of adverse events. Adverse events diminish or disappear after stopping using tested products, and symptoms occur once again with the use of tested products.

9.7 report and record: ①serious adverse events: clinical safety management must be informed by fax or scaning within 24 hours, regardless of whether the event is related to the tested product. When it's the first time to report, or each time when SAE needs modification, researchers need to complete serious adverse events spreadsheet in the eCRF, The spreadsheet will be automaticly sent to clinical safety manager xt211311@aliyun.com in the form of email. All serious adverse events are also required in the eCRF spreadsheet severity column to choose "serious". ②Not serious adverse events: all not serious adverse events must be recorded on the eCRF's adverse events page.

9.8 follow-up visits: All serious adverse events should be followed up until the outcome of the event. The researchers need to inform the clinical safety manager of any follow-up information within 24 hours, such as changes in diagnosis, results, the date of remission, the termination of treatment, and so on.

If serious adverse events persist after discontinuation of the study, follow-up is required. In addition, when adverse events occur, if it's necessary to further evaluate the causal relationship between adverse events and the tested product, then all the examinations and laboratory results must be recorded in the case report form or attached document. Within 30 days after the last use of the study product, the SAE also needs to be reported in the same way within 24 hours.

9.9 Inform: The sponsor is responsible for the safety evaluation of the tested product. The sponsor must promptly inform all researchers, observational hospitals and regulatory authorities of any discoveries that are likely to affect subjects' safety, influence study process, change the ethics committee's attitude to approve or agree that research continues.

9.10 Report: The sponsor must accelerate reporting to all investigators, observational hospitals, IRB (S) /IEC (s) and management authorities (if necessary) about all serious and suspicious unexpected serious adverse reactions (SUSAR).

This accelerated report needs to comply with applicable regulatory requirements, and ICH guidelines on the management of clinical safety data: standards of accelerated reporting.

The sponsor should submit all latest progress and staged reports of security to management authorities, according to applicable regulatory requirements

ELIGIBILITY:
Inclusion Criteria:

* 1 to 2 months-old term infants (gestational age ≥37 weeks) checked-up in child care department
* Gender not limited
* Though completely understanding the importance of breast milk feeding, subjects' mothers cann't continue to give breast milk feeding owing to their own problems, and have to feed infants with foumula milk only
* Legal guardians of subjects know the objective of this study and get the tested formula milk for free, then volunteer to participate in the study and sign an informed consent

Exclusion Criteria:

* Infants' mothers suffered from infectious diseases during pregnancy
* Subjects suffered from basic diseases (such as congenital heart disease and genetic metabolic diseases) and congenital deformity
* Brain damage caused by a variety of factors such as HIE, intraventricular hemorrhage, hypoglycemia
* Small for gestational age
* Subjects cann't get full enteral feeding, such as NEC
* Subjects allergic to cow's milk protein
* Subjects used antibiotics before inclusion
* Subjects participate in other clinical trials before inclusion or during this trial

Drop-out Criteria:

* Subjects in violation of this trial plan (using the other brand formula or not according to the plan)
* Loss of follow-up
* Withdrawing the informed consent or asked to quit on their own

Ages: 4 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 216 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Growth rate of height | At the end of 12 weeks after feeding
  (The height at the end of 12 weeks after feeding minus the height before feeding)/3
Growth rate of weight | At the end of 12 weeks after feeding
  (The weight at the end of 12 weeks after feeding minus the weight before feeding)/3
Growth rate of head circumference | At the end of 12 weeks after feeding
  (The head circumference at the end of 12 weeks after feeding minus the head circumference before feeding)/3

SECONDARY OUTCOMES:
Growth rate of height | At the end of 4 weeks after feeding
  (The height at the end of 12 weeks after feeding minus the height before feeding)/1
Growth rate of height | At the end of 8 weeks after feeding
  (The height at the end of 12 weeks after feeding minus the height before feeding)/2
Growth rate of weight | At the end of 4 weeks after feeding
  (The weight at the end of 12 weeks after feeding minus the weight before feeding)/1
Growth rate of weight | At the end of 8 weeks after feeding
  (The weight at the end of 12 weeks after feeding minus the weight before feeding)/2
Growth rate of head circumference | At the end of 4 weeks after feeding
  (The head circumference at the end of 12 weeks after feeding minus the head circumference before feeding)/1
Growth rate of head circumference | At the end of 8 weeks after feeding
  (The head circumference at the end of 12 weeks after feeding minus the head circumference before feeding)/2
Defecate frequency | At the end of 4 weeks after feeding
  Evaluated by subjects' guardians
Defecate frequency | At the end of 8 weeks after feeding
  Evaluated by subjects' guardians
Defecate frequency | At the end of 12 weeks after feeding
  Evaluated by subjects' guardians
Fresh stool character | At the end of 4 weeks after feeding
  Fresh stool (collect stool data over 3 days) character at the end of 4 weeks, evaluated by Bristol stool shape chart and divided into 7 type, the subjects' guardians need to record it and call to child care doctor
Fresh stool character | At the end of 8 weeks after feeding
  Fresh stool (collect stool data over 3 days) character at the end of 8 weeks, evaluated by Bristol stool shape chart and divided into 7 type, the subjects' guardians need to record it and call to child care doctor
Fresh stool character | At the end of 12 weeks after feeding
  Fresh stool (collect stool data over 3 days) character at the end of 12 weeks, evaluated by Bristol stool shape chart and divided into 7 type, the subjects' guardians need to record it and call to child care doctor
Eye secretions | After waking up at the end of 4 weeks after feeding
  The subjects' guardian needs to take photos of eye secretions and send photos to research Centre, evaluated by specialists
Eye secretions | After waking up at the end of 8 weeks after feeding
  The subjects' guardian needs to take photos of eye secretions and send photos to research Centre, evaluated by specialists
Eye secretions | After waking up at the end of 12 weeks after feeding
  The subjects' guardian needs to take photos of eye secretions and send photos to research Centre, evaluated by specialists

CONTACTS AND LOCATIONS:
Overall Officials: Chongfan Zhang, Bachelor, Study Director — Children's Hospital of Fudan University; Wei Xiang, Master, Principal Investigator — Maternal and Child Health Hospital of Hainan Province
Locations (6):
- China (6):
  - Z1, Zhangzhou, Fujian
  - Z2, Zhangzhou, Fujian
  - H2, Haikou, Hainan
  - H1, Haikou, Hainan
  - BJ1, Baoji, Shanxi
  - BJ2, Baoji, Shanxi

IPD SHARING:
Plan to Share IPD: Yes